CLINICAL TRIAL: NCT04121442
Title: Phase I/IIa, Non-Randomised, Open-Label Dose Escalation and Expansion Trial With Isunakinra Alone and in Combination With a PD-1/PD-L1 Inhibitor in Patients With Metastatic or Unresectable, Locally Advanced Malignant Solid Tumors
Brief Title: Isunakinra Alone and in Combination With a PD-1/PD-L1 Inhibitor in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Buzzard Pharmaceuticals (Industry)
Collaborators: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BUZ01CD101
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — EBI-005

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Isunakinra monotherapy and in combination w PD-(L)1 Inhibitor (Experimental): Patients will receive specified dose of Isunakinra as monotherapy for three weeks, followed by combination with a PD-(L)1 inhibitor
  Interventions: Biological: Isunakinra; Biological: PD-(L)1 Inhibitor

INTERVENTIONS:
Biological: Isunakinra — Isunakinra is a recombinant protein that binds to the IL1R1 and potently blocks IL-1 alpha and IL-1 beta signaling
  Other Names: EBI-005
Biological: PD-(L)1 Inhibitor — Monoclonal antibody targeting PD-1 or PD-L1

SUMMARY:
Isunakinra - a potent Interleukin-1 receptor inhibitor - will be given to patients with solid tumors to determine safety and tolerability of three different doses. Isunakinra will then be combined with a PD-(L)1 inhibitor. Pharmacokinetics and Pharmacodynamic effects of monotherapy treatment as well as the combination will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have:

   * Metastatic or unresectable locally advanced malignant solid tumor.
   * Histologic confirmation.
2. The study patients are required to have measurable disease by radiographic criteria (RECIST 1.1) and irRC.
3. Prior therapy: Patients must have completed or had disease progression on at least one prior line of disease-appropriate therapy for metastatic disease (with or without PD-1 inhibitors), with no available therapy likely to convey clinical benefit, or not be candidates for therapy of proven efficacy for their disease.
4. There should be a minimum of 2 weeks from any prior chemotherapy, immunotherapy and/or radiation and 4 weeks washout period for immunotherapy. Patients with prostate cancer on hormone deprivation therapy may continue that therapy while on study.
5. Patients must have recovered (grade 1 or baseline) from any clinically significant toxicity associated with prior therapy (for example, alopecia is not clinically significant). Typically, this approximates 3-4 weeks for patients who most recently received cytotoxic therapy, except for the nitrosoureas and mitomycin C, for which 6 weeks is needed for recovery.
6. Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of this agent in patients < 18 years of age, children are excluded from this study but will be eligible for future pediatric trials.
7. ECOG performance status ≤ 1
8. Patients must have normal organ and hematologic function as defined below:

   * Serum creatinine ≤ 1.5 x upper limit of normal OR creatinine clearance and a 24-h urine collection of ≥ 60 mL/min.
   * ALT and AST ≤ 3x the upper limits of normal.
   * Total bilirubin ≤ 1.5 x upper limit of normal OR in patients with Gilbert's syndrome, a total bilirubin ≤ 3.0.
   * Hematological eligibility parameters (within 16 days of starting therapy):

     * Granulocyte count ≥ 1,500/mm3
     * Platelet count ≥ 75.000/mm3
9. Patients must have baseline pulse oximetry > 90% on room air.

Exclusion Criteria:

1. Pregnant women or women presently breast-feeding their children are excluded due to unknown risks to a developing fetus or infant, confirmed by negative pre-treatment serum pregnancy test.
2. Concurrent treatment for cancer, with specific exceptions noted in inclusion criteria.
3. Any significant disease that, in the opinion of the investigator, may impair the patient's tolerance of study treatment.
4. Significant dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
5. Active autoimmune diseases requiring treatment. However, patients with vitiligo, alopecia, or clinically stable autoimmune endocrine disease who are on appropriate replacement therapy (if such therapy is indicated) are eligible.
6. Concurrent use of systemic steroids, except for physiologic doses of systemic steroid replacement or local (topical, nasal, or inhaled) steroid use. Limited pharmacologic doses of systemic steroids (e.g., in patients with exacerbations of reactive airway disease or to prevent iv contrast allergic reaction or anaphylaxis in patients who have known contrast allergies) are allowed.
7. Patients who are receiving any other investigational agents within 28 days before start of study treatment.
8. Patients with untreated central nervous system metastases or local treatment of brain metastases within the last 6 months. Patients with stable brain metastasis for 6 months post-intervention are eligible.
9. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the agents used in study.
10. Serious or uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
11. HIV-positive patients are ineligible because of the potential for decreased immune response.
12. Patients unwilling to use adequate contraception (defined as hormonal or barrier method or abstinence) prior to study entry are excluded. If the patient needs to be on adequate contraception, contraception must start before study entry and continue for 3 months after completion of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who experience DLTs | From baseline to 49 days of treatment
  The primary endpoint of this study is the proportion of patients who experience DLTs. The MTD (Maximum Tolerated Dose) will be determined based on the dose escalation cohorts. The evaluation period for DLTs will be 21 days following the first dose of Isunakinra and 28 days following addition of PD1-PDL1 inhibitor
Proportion of patients who experience decrease of IL-6 or hsCRP by >20% | From baseline to 49 days of treatment
  Optimal Biological Dose (OBD) as indicated by changes in IL-6 and hsCRP plasma levels.

SECONDARY OUTCOMES:
Percent of individuals who experience radiographic response | Two years
  Overall response rate (ORR) by RECIST 1.1
Progression-free survival (PFS) | Two years
  Defined as the time, in days, between treatment initiation and when the patient is found to have recurrent and/or metastatic disease on imaging, or death for any reason.
Overall survival | Two years
  Defined as the time, in days, between treatment initiation and when the patient dies from any cause regardless of etiology.

CONTACTS AND LOCATIONS:
Overall Officials: Maarten de Chateau, MD, PhD, Study Director — Buzzard Pharmaceuticals
Locations (1):
- Baylor Charles A. Simmons Cancer Center, Dallas, Texas, United States

REFERENCES:
- [Background] Hou J, Townson SA, Kovalchin JT, Masci A, Kiner O, Shu Y, King BM, Schirmer E, Golden K, Thomas C, Garcia KC, Zarbis-Papastoitsis G, Furfine ES, Barnes TM. Design of a superior cytokine antagonist for topical ophthalmic use. Proc Natl Acad Sci U S A. 2013 Mar 5;110(10):3913-8. doi: 10.1073/pnas.1217996110. Epub 2013 Feb 19. PMID 23431173
- [Background] Kovalchin J, King B, Masci A, Hopkins E, Fry J, Hou J, Li C, Tenneson K, Weber S, Wolfe G, Collins K, Furfine ES. Preclinical Development of EBI-005: An IL-1 Receptor-1 Inhibitor for the Topical Ocular Treatment of Ocular Surface Inflammatory Diseases. Eye Contact Lens. 2018 May;44(3):170-181. doi: 10.1097/ICL.0000000000000414. PMID 28727604
- See also: Hou et al PNAS 2013 Generation and Characterisation of Isunakinra — https://www.ncbi.nlm.nih.gov/pubmed/23431173
- See also: Kovalchin et al Eye Contact Lens 2018. Pre-clinical Characterisation of Isunakinra — https://www.ncbi.nlm.nih.gov/pubmed/28727604